CLINICAL TRIAL: NCT06691737
Title: Effect of Whole-body Vibration on Postural Stability, Muscle Flexibility and Lower Limb Power in Young Basketball Players with Generalized Joint Hypermobility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AWFiS/2024_4_OF
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Generalized Joint Hypermobility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Generalized Joint Hypermobility (Experimental)
  Interventions: Other: Whole Body Vibration
- Not Generalized Joint Hypermobility (Experimental)
  Interventions: Other: Whole Body Vibration

INTERVENTIONS:
Other: Whole Body Vibration — Whole body vibration consists of 3-minute vibrations with a 30-second break. Participants were asked to step onto the platform barefoot and position their feet "3" from the center of the platform, with feet pointing forward, knees slightly bent, and upper limbs along the body. The training was divided into two parts: week 1 with a frequency of 20 Hz, and a constant amplitude of 3 mm.

SUMMARY:
The goal of this clinical trial is to assess the effect of whole body vibration (WBV) on postural stability, flexibility of the lumbar-pelvic-hip complex and lower leg muscles, and jumping ability in basketball players aged 9-15 years. The main questions it aims to answer are:

Does WBV affect the level of postural stability in basketball players aged 9-15 years? Does WBV affect the level of postural stability in basketball players aged 9-15 years? Does WBV affect the flexibility of the iliopsoas, rectus femoris, posterior group of hamstrings, soleus and gastrocnemius in basketball players aged 9-15 years? Does WBV affect the jump height, relative peak power, contraction time in basketball players aged 9-15 years?

Participants will take part in 6 vibration sessions at 20Hz over 6 weeks. Vibration will be performed on the Galileo Med35 platform (3x3 min).

ELIGIBILITY:
Inclusion Criteria:

* Men aged 9-15
* Playing basketball in a sports club at least 2 training sessions a week

Exclusion Criteria:

* Thrombosis (acute narrowing of blood vessels),
* Inflammation of the musculoskeletal system,
* Arthropathy,
* Hernias,
* Discopathies,
* Tendonitis,
* Fresh fractures,
* Scars,
* Surgeries,
* Kidney stones,
* Rheumatoid arthritis,
* Implants in the body,
* Epilepsy,
* Current injuries to the musculoskeletal system,
* Occurrence of chronic pain complaints of the musculoskeletal system.

Ages: 9 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-06-04 (Estimated)

PRIMARY OUTCOMES:
Changes in Postural Stability | 6 weeks before the intervention, the day before the intervention began, the day after the intervention, and 6 weeks after the intervention.
  Postural stability was measured as the overall stability index (OSI) on the Biodex Balance System on the stable and unstable platform with open and closed eyes.
Range of motion (ROM) of the ankle, knee, and hip joints. | 6 weeks before the intervention, the day before the intervention began, the day after the intervention, and 6 weeks after the intervention.
  Range of motion (ROM) of the ankle, knee, and hip joints, will be measured in a resting position using an inclinometer for the iliopsoas, rectus femoris, posterior hamstring, soleus, and gastrocnemius muscles separately.
Countermovement Jump Performance | 6 weeks before the intervention, the day before the intervention began, the day after the intervention, and 6 weeks after the intervention.
  Countermovement jump performance will be measured by using force plates, It will be assessed Jump height (JH), relative peak power (RPP), and contraction time (CT).